CLINICAL TRIAL: NCT05326217
Title: The Effects of Exercise and Probiotics on the Efficacy and Possible Mechanisms of Dysmenorrhea From the Perspective of Microbiome
Brief Title: The Effects of Exercise and Probiotics on Dysmenorrhea and Microbiome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Principal Investigator, Wen Ching Huang, Associated professor, National Taipei University of Nursing and Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FJU-IRB-C110039
Record Dates: First submitted 2022-03-29; First posted 2022-04-13 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Dysmenorrhea; Inflammation; Microbial Substitution
Keywords: Lactobacillus; Sport nutrition
MeSH Terms: conditions — Dysmenorrhea; Inflammation | interventions — Exercise

STUDY DESIGN:
Masking Description: First stage: Open Label Second stage: Single Blind for probiotics treatment
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control Group (No Intervention): non-dysmenorrhea population with original lifestyle
- Dysmenorrhea (No Intervention): dysmenorrhea population without exercise intervention
- Dysmenorrhea+Aerobic Exercise (Experimental): dysmenorrhea population with aerobic exercise intervention
  Interventions: Other: Aerobic exercise
- Dysmenorrhea+Resistant Exercise (Experimental): dysmenorrhea population with resistant exercise intervention
  Interventions: Other: Resistant exercise

INTERVENTIONS:
Other: Aerobic exercise — The aerobic exercise :In this study, the exercise intensity is set based on the subject's maximum heart rate, and the target heart rate is adjusted according to the literature to reach 60-90% of the maximum heart rate. A gradual increase of intermittent exercise will be designed for current exercise prescription. In terms of exercise frequency and time, there will be two times interventions per week for at least 60 minutes per time (including warm-up and cool down exercises).
  Arms: Dysmenorrhea+Aerobic Exercise
Other: Resistant exercise — The resistant exercise : muscular endurance (15-20RM) and muscular hypertrophy (8-12RM) are applied to main exercise intensity. The intensity is gradually adjusted according to the state of each subject, and the intervention is performed twice a week (50 minutes per time).The target muscles of resistance training include quadriceps femoris, biceps femoris, calf muscles, core muscles (including pelvic floor muscles), back muscles, pectoralis major, biceps/triceps and other muscle groups.
  Arms: Dysmenorrhea+Resistant Exercise

SUMMARY:
The study try to investigate the possible effects of exercise and probiotics supplementation on dysmenorrhea amelioration from the perspective of microbiome.

DETAILED DESCRIPTION:
In current study, there were two stages designed for current study. The definition of dysmenorrhea population depended on the Visual Analogue Scale (VAS) of McGill Pain Questionnaire (more than 5) and the VAS score less than 2 was considered as non-dysmenorrhea population.

In the first stage, the 20 subjects were recruit for non-dysmenorrhea group (Control group) and other 60 subjects were randomly allocated into three group with original lifestyle, aerobic, and resistant exercise intervention (Dys-Control, Dys-Aerobic, and Dys-resistant groups). The questionnaires (Premenstrual syndrome, the Menstrual Distress, and McGill Pain), body composition, physical fitness, biochemistries, inflammation, hormones and microbiome analysis (feces and tampon) were evaluated and assessed before and after 10-weeks indicated exercise training.

In the second stage, one hundred subjects (20 non-dysmenorrhea and 80 dysmenorrhea populations) will be recruited and the dysmenorrhea will be randomly allocated into Dys-Control, Dys-probiotics, Dys-exercise and Dys-probiotics and exercise groups. The questionnaires (Premenstrual syndrome, the Menstrual Distress, and McGill Pain), body composition, physical fitness, biochemistries, inflammation, hormones and microbiome analysis (feces and tampon) were evaluated and assessed before and after 10-weeks indicated interventions (probiotics and exercise).

ELIGIBILITY:
Inclusion Criteria:

* Primary dysmenorrhea
* Visual Analog Score of McGill pain questionnaire (0-2 for non-dysmenorrhea; >5 for dysmenorrhea)

Exclusion Criteria:

* Pregnancy, menstrual disorders, obesity (BMI>30), smoking, and alcohol or drug addiction
* Cardiovascular disease, hypertension, diabetes, asthma, chronic pulmonary obstruction, mental illness

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-01-20 (Actual); Primary Completion 2023-01-19 (Estimated); Study Completion 2023-01-19 (Estimated)

PRIMARY OUTCOMES:
The effects of different types of exercise on premenstrual syndrome questionnaire with dysmenorrhea | 10 weeks
  The premenstrual syndrome questionnaire is applied for evaluation of premenstrual syndromes before mense. A higher score indicates severer indicated syndromes. Changes of the premenstrual syndrome questionnaire measure will be assessed at the 0 week and 10 weeks.
The effects of different types of exercise on menstrual distress questionnaire with dysmenorrhea | 10 weeks
  The menstrual distress questionnaire is applied for evaluation of distress syndromes during mense. A higher score indicates severer indicated syndromes. Changes of the menstrual distress questionnaire measure will be assessed at the 0 week and 10 weeks.
The effects of different types of exercise on McGill pain questionnaire with dysmenorrhea | 10 weeks
  The McGill pain questionnaire is applied for evaluation of types and degrees of pain during mense. A higher score indicates severer indicated syndromes. Changes of theMcGill pain questionnaire measure will be assessed at the 0 week and 10 weeks.
The effects of different types of exercise on cardiovascular capacity | 10 weeks
  The cardiovascular capacity is evaluated by 3-minute step test. The higher index of cardiovascular capacity means the higher cardiovascular fitness. Changes of cardiovascular capacity will be assessed at the 0 week, and 10 weeks.
The effects of different types of exercise on muscular strength of upper limbs | 10 weeks
  The muscular strength of upper limbs is evaluated by grip-strength test. The higher strength of test means the higher strength fitness in upper limbs. Changes of muscular strength of upper limbs will be assessed at the 0 week, and 10 weeks.
The effects of different types of exercise on power | 10 weeks
  The power is evaluated by standing long jump. The higher distance of test means the higher power fitness. Changes of power will be assessed at the 0 week, and 10 weeks.
The effects of different types of exercise on core strength | 10 weeks
  The core strength endurance is evaluated by 1-minute bent-knee sit-up test. The higher repetitions mean the higher core strength endurance fitness. Changes of core strength endurance will be assessed at the 0 week, and 10 weeks.
The effects of different types of exercise on body composition | 10 weeks
  The body composition was simultaneously measured by Inbody 270 (Bioelectrical Impedance Analysis) for outcome measures including body-fat percentage, and muscular percentage in the upper and lower limbs. The higher muscular percentage and lower body-fat percentage are associated with better fitness. Changes of body-fat percentage, and muscular percentage in the upper and lower limbs measures will be assessed at the 0 week, and 10 weeks.
The microbiome succession of the dysmenorrhea with different types of exercise intervention | 10 weeks
  Determination of the gut microbiota composition from the feces and tampon samples by 16S metagenomic, data analysis and building of a mathematical model to test the potential modulation of the gut microbiota architecture for primary dysmenorrhea.Changes of microbiota succession in the feces and tampons will be assessed at the 0 week, and 10 weeks.
The effects of different types of exercise on cytokines in dysmenorrhea | 10 weeks
  The cytokines was simultaneously measured by enzyme-linked immunosorbent assay for outcome measures including TNF-α, IL-1β, IL-6, and IL-10. The higher TNF-α, IL-1β, and IL-6 cytokines mean the higher inflammation and higher IL-10 mean the higher immunosuppression. Changes of cytokines measures will be assessed at the 0 week, and 10 weeks.
The effects of different types of exercise on biochemistries in dysmenorrhea | 10 weeks
  The biochemical variables were simultaneously measured by automated clinical chemistry analyzer for outcome measures including VEGF, Estrogen, Progesterone, adrenaline, cortisol, serotonin, PEG2, PGF2α, Prostacyclin, and Thromboxane. The expressive levels of indicated indexes mean different physiological modulations. Changes of biochemical measures will be assessed at the 0 week, and 10 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Wen Ching Huang, PhD, Principal Investigator — National Taipei University of Nursing and Health Sciences
Locations (1):
- National Taipei University of Nursing and Health Sciences, Taipei, Taiwan